CLINICAL TRIAL: NCT02980107
Title: Presenting Summary Information From Cochrane Systematic Reviews: Protocol for Research of Infographics Presentation vs. Plain Language Summary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Split (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Principal Investigator, Ivan Buljan, Research Assistant, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IP-2014-11-7672
Record Dates: First submitted 2016-11-25; First posted 2016-12-02 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLS (Active Comparator): The control group will receive PLS: text format with simple explanation of the survey topic main findings and is intended for lay audience.
  Interventions: Other: PLS
- Infographics (Experimental): Infographics format of a Cochrane systematic review summary represents the experimental intervention in the trial, where the results are presented with text and pictures.
  Interventions: Other: Infographics

INTERVENTIONS:
Other: Infographics — Cochrane started developing infographics, where short textual information about research is supported by visual representations of the main findings and is also aimed at the lay public The investigators will examine whether this format is better in information uptake than standard PLS.
  Arms: Infographics
Other: PLS — Text format with simple explanation of the survey topic main findings and is intended for lay audience.
  Arms: PLS

SUMMARY:
The objective of this study is to evaluate the efficacy of infographics, compared to standard PLS format, in presenting information, in terms of understanding and remembering research results by consumers.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) with two different formats of the same systematic review summary (Infographics, PLS). The content of these two formats is based on the same systematic review, but the ways of data presentation will differ: visual presentation in plain language and plain language only. The interventions will be delivered online in November 2016, with members of the consumers' groups for pregnancy and parenting - RODA ("Roditelji u akciji", engl."Parents in action"), which gathers different types of consumers: pregnant women, young mothers and parenting and pregnancy advisors; and the members of the Association for Patients' Rights. The trial will be voluntary and anonymous. The survey will consist of 5 parts, in the following order: 1) one format of the summary (randomly assigned), 2) health numeracy, 3) demographic data 4) comprehension test of the information given in the summary, and 5) user friendliness of information and overall satisfaction with the given summary assessed by survey.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be members of RODA and Association for Patients' Rights (women) .

Exclusion Criteria:

* Male members of RODA and Association for Patient's Rights

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Buljan, Principal Investigator — Researcher
Locations (1):
- University of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Osborn CY, Wallston KA, Shpigel A, Cavanaugh K, Kripalani S, Rothman RL. Development and validation of the General Health Numeracy Test (GHNT). Patient Educ Couns. 2013 Jun;91(3):350-6. doi: 10.1016/j.pec.2013.01.001. Epub 2013 Feb 21. PMID 23433635
- See also: Web page where new formats for presentation of Cochrane systematic reviews can be found. — http://visuallycochrane.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Plain Language Summary: The control group will receive PLS: text format with simple explanation of the survey topic main findings and is intended for lay audience.
  PLS: Text format with simple explanation of the survey topic main findings and is intended for lay audience.
Period: Overall Study
Arm/Group | Plain Language Summary | Infographics
Started | 105 | 107
Completed | 54 | 45
Not Completed | 51 | 62
Not completed — Withdrawal by Subject | 51 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Language Summary | Infographics | Total
Number analyzed (Participants) | 54 | 45 | 99
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [32 to 40] | 37 [32 to 42] | 38 [32 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 45 | 99
  Male | 0 | 0 | 0
Heard of Cochrane systematic reviews [Count of Participants; unit: Participants] | 23 | 25 | 48
Used Cochrane library [Count of Participants; unit: Participants] | 12 | 16 | 28
Primary source of health information [Count of Participants; unit: Participants]
  Internet | 33 | 33 | 66
  Family Members | 4 | 0 | 4
  Family physician | 12 | 5 | 17
  Library | 2 | 1 | 3
  Other | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Understanding of the Summary Content
Description: The questions will focus on understanding the benefits and risks of the intervention and the quality of evidence described in the systematic review. There will be 10 open ended questions, which will be assessed by two assessors, and the total score will be the sum of correct answers (total score ranging from 0-10). Higher scores would represent greater understanding of the content.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics
Number analyzed (Participants) | 54 | 45
units on a scale | 7.0 [6.0 to 7.0] | 7.0 [6.0 to 7.0]

2. Secondary Outcome: Reading Experience
Description: This section of the survey will include 5 questions about the experience of participants about the text they read, measured on a 10-point Likert type scale, where 1 means do not agree at all and 10 means fully agree. The total score is the sum of scores on all five answers (minimum 5, maximum 50). Greater scores indicate more positive reading experience.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics
Number analyzed (Participants) | 54 | 45
units on a scale | 22.5 [19.0 to 27.4] | 33.0 [28.0 to 36.0]

3. Secondary Outcome: User Friendliness
Description: This section of the survey will have 5 questions concerning how easy it was for the participant to find relevant information, measured by a 10-point Likert type scale where the answer 1 means I do not agree at all and 10 means I fully agree. The total score is the sum of scores on all the answers (minimum 5, maximum 50). Higher scores indicate greater perception of the summary format as more user friendly.
Time Frame: One month (30 days)
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics
Number analyzed (Participants) | 54 | 45
units on a scale | 21.0 [19.0 to 25.0] | 30.0 [25.5 to 34.5]

4. Other Pre Specified Outcome: Health Numeracy
Description: This section will use 6-item General health numeracy test (Osborne et al., 2013) in order to determine how much our participants understand the basic health instructions regarding numeracy dimension. For each correct answer, the participants receive one point and the total score is the sum of all correct answers.
Time Frame: One month (30 days)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Plain Language Summary | Infographics
Number analyzed (Participants) | 54 | 45
units on a scale | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 5.0]

ADVERSE EVENTS:
Time Frame: No adverse events were collected.
Description: 0
Arm/Group | Plain Language Summary | Infographics
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor had no role in the research planning, its execution nor publication.